CLINICAL TRIAL: NCT01288105
Title: Use of Optical Coherence Tomography to Determine the Optimal Management of Patients With Drug-eluting Stents Who Need Non-cardiac Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Teresa D. Moore, IRB administrator, VA North Texas Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 10-106
Record Dates: First submitted 2011-01-20; First posted 2011-02-02 (Estimated); Last update posted 2011-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Coronary Stent Occlusion
Keywords: drug-eluting stents; noncardiac surgery
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Optical Coherence Tomography (Experimental): Patients enrolled in the study will undergo optical coherence tomography to evaluate the extent of stent strut coverage.
  Interventions: Device: Optical coherence tomography

INTERVENTIONS:
Device: Optical coherence tomography — Optical coherence tomography will be performed to determine the stent strut coverage. Patients in whom >95% of stent struts are covered will not receive perioperative bridging with a glycoprotein IIb/IIIa inhibitors, whereas those with <95% stent strut coverage will receive perioperative bridging.
  Other Names: invasive intracoronary imaging

SUMMARY:
The specific aim of this proposal is to examine the impact of OCT and IVUS-guided management of patients with prior DES implantation who need major non-cardiac surgery and discontinuation of dual antiplatelet therapy on the perioperative (1 week prior to surgery until 30 days post surgery) incidence of major adverse cardiac events.

DETAILED DESCRIPTION:
Patients who receive drug-eluting stents (DES) and subsequently require non-cardiac surgery have increased risk for perioperative stent thrombosis, especially when antiplatelet therapy discontinuation is required. Perioperative administration of a glycoprotein IIb/IIIa inhibitor may decrease the stent thrombosis risk, but it is cumbersome and carries high cost. Stents that have been endothelialized by optical coherence tomography (OCT) are likely to have low risk for perioperative stent thrombosis and therefore intensive management strategies, such as "bridging with a glycoprotein IIb/IIIa inhibitor" would not be required. The current study will assess whether OCT utilization can help optimize the preoperative management of DES patients requiring major non-cardiac surgery.

The specific aim of this proposal is to examine the impact of OCT and IVUS-guided management of patients with prior DES implantation who need major non-cardiac surgery and discontinuation of dual antiplatelet therapy on the perioperative (1 week prior to surgery until 30 days post surgery) incidence of major adverse cardiac events.

The hypothesis is that OCT and IVUS-guided treatment will have low incidence (≤10%) of perioperative major adverse cardiac events.

The specific aim of this proposal is to examine the impact of OCT and IVUS-guided management of patients with prior DES implantation who need major non-cardiac surgery and discontinuation of dual antiplatelet therapy on the perioperative (1 week prior to surgery until 30 days post surgery) incidence of major adverse cardiac events.

The hypothesis is that OCT and IVUS-guided treatment will have low incidence (≤10%) of perioperative major adverse cardiac events.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Need for major non-cardiac surgery requiring discontinuation of dual antiplatelet therapy
* Agree to participate and provide informed consent

Exclusion Criteria:

* Patients who have a creatinine above 2.5 mg/dL (unless they require hemodialysis, in which case they are eligible to participate)
* Challenging vascular access
* History of an allergic reaction to glycoprotein IIb/IIIa inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 30-days post surgery
  composite of cardiac death, myocardial infarction, coronary revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S Brilakis, MD, PhD, Principal Investigator — North Texas Veterans Healthcare System
Locations (1):
- VA North Texas Healthcare System, Dallas, Texas, United States